CLINICAL TRIAL: NCT03410719
Title: Effectiveness of Pasta and Other Starchy Foods With a Low Glycemic Response to Promote Cardio-metabolic and Emotional Well-being.
Brief Title: Mediterranean Style Diet and Low Glycemic Responses
Acronym: MedGICarb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Federico II University (Other); University of Agriculture Science, Uppsala, Sweden (Unknown)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16100183
Record Dates: First submitted 2018-01-11; First posted 2018-01-25 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: block randomized, parallel, controlled,
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- <55 (Low-GI group) (Experimental): intervention weeks 1-12 the subjects in each group will be counseled to follow their weight maintaining assigned diet using a combination of prescribed menus (breakfast, lunch, and snack eating occasions) and an item specific version of the Pasta Recipe Builder (dinner). The two group-specific diet plans will mostly contain the same foods and beverages typically included in Mediterranean-style diets, except for substitutions of major sources of carbohydrate in their meals:Low-GI - pasta, barley, parboiled rice, legumes.
  Interventions: Other: Hi GI
- >70 (Hi-GI group). (Experimental): intervention weeks 1-12 the subjects in each group will be counseled to follow their weight maintaining assigned diet using a combination of prescribed menus (breakfast, lunch, and snack eating occasions) and an item specific version of the Pasta Recipe Builder (dinner). The two group-specific diet plans will mostly contain the same foods and beverages typically included in Mediterranean-style diets, except for substitutions of major sources of carbohydrate in their meals: Hi-GI - rice, potato,
  Interventions: Other: Hi GI

INTERVENTIONS:
Other: Hi GI — subjects will consume the same quantities of metabolizable CHOs (270 g/d) with 135 g of CHOs assigned to the GI intervention foods. The 135 g of CHOs will be distributed as 35 g GI breakfast product, 40 g GI lunch product, and 60 g GI dinner product. Assuming an average 2400 kcal/d total energy requirement among subjects, the 270 g/d metabolizable CHO equates to 40% of total energy intake (1080 kcal/d). One-half of daily CHO intake (135 g/d) will be the same between the Hi-GI and Low-GI groups, including CHOs in fruits, vegetables, and other foods that all subjects will consume. The other one-half of daily CHO intake (135 g) will be different between the Low-GI and Hi-GI groups. Specifically, the GI values of these foods will either be <55 (Low-GI group) or >70 (Hi-GI group).
  Other Names: Low GI

SUMMARY:
the aim of this study is to evaluate whether a Mediterranean diet rich in pasta and other starchy foods with a (Low-GI), as compared with a similar Mediterranean diet containing very little pasta and based on starchy foods with a (Hi-GI) is able to reduce insulin and glucose concentrations during a prolonged test study meal.

DETAILED DESCRIPTION:
The overall aim of this study is to evaluate whether a Mediterranean diet rich in pasta and other starchy foods with a low glycemic response (Low-GI), as compared with a similar Mediterranean diet containing very little pasta and based on starchy foods with a high glycemic response (Hi-GI) is able to reduce insulin and glucose concentrations during a prolonged test study meal.

ELIGIBILITY:
Inclusion Criteria:

* • BMI 25-37 kg/m2 with a waist circumference > 102 cm (males) or > 88 cm (females) and one additional feature of Metabolic Syndrome according to ATPIII [1], including blood pressure > 130/85 or treatment, fasting plasma glucose >100mg/dL, fasting triglycerides >150 mg/dL, HDL cholesterol < 40 mg/dL (males) or 50 mg/dL (females),

  * weight stable (± 3 kg in previous 3 mo);
  * no acute illness; and non-diabetic.

Exclusion Criteria:

* age <30 and >69years;
* fasting triglycerides ≥400 mg/dL;
* fasting cholesterol >240 mg/dL or low-density lipoprotein cholesterol>160 mg/dL
* fasting glucose >126 mg/dL,
* systolic blood pressure >160 mmHg, diastolic blood pressure >100 mmHg
* a BMI >37 kg/m2, weight changes during the previous 3 months (greater than ± 3 kg),
* stable intensive physical activity regimen during the previous 3 months (>3 h/wk of moderate or high intensity exercise, resistance or aerobic training).
* cardiovascular events (myocardial infarction or stroke) during the 6 months prior to the study;
* renal and liver failure (creatinine >1.7 mg/dl and ALT/AST >2 times than normal values, respectively);
* anaemia (Hb <12 g/dL);
* diabetes mellitus.
* If you are pregnant

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
The effects of Low-GI and Hi-GI diets | 15weeks
  All subjects will consume the same quantities of metabolizable carbohydrate (270 g/d) with 135 g of carbohydrates assigned to the GI intervention foods. The 135 g of carbohydrates will be distributed as 35 g GI breakfast product, 40 g GI lunch product, and 60 g GI dinner product. Fiber is set as 35 g/d for both intervention groups. Assuming an average 2400 kcal/d total energy requirement among subjects, the 270 g/d metabolizable CHO equates to 40% of total energy intake (1080 kcal/d). One-half of daily CHO intake (135 g/d) will be the same between the Hi-GI and Low-GI groups, including CHOs in fruits, vegetables, and other foods that all subjects will consume. The other one-half of daily CHO intake (135 g) will be different between the Low-GI and Hi-GI groups. Specifically, the GI values of these foods will either be <55 (Low-GI group) or >70 (Hi-GI group).

SECONDARY OUTCOMES:
Insulin Sensitivity | 15 weeks
  Measures of Insulin Sensitivity will include fasting serum lipid-lipoprotein profile, plasma fasting and postprandial glucose, insulin, CRP, C-peptide, fasting HbA1c, 24-hour interstitial continuous glucose monitoring (Medtronic ipro2 Professional CGM device (Northridge, CA).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Riccardi (riccardi@unina.it), M.D, Principal Investigator — Federico II University; Rikard Landberg (rikard.landberg@slu.), Ph.D, Principal Investigator — Uppsala University, Uppsala, Sweden
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giosue A, Skantze V, Hjorth T, Hjort A, Brunius C, Giacco R, Costabile G, Vitale M, Wallman M, Jirstrand M, Bergia R, Campbell WW, Riccardi G, Landberg R. Association of the glucose patterns after a single nonstandardized meal with the habitual diet composition and features of the daily glucose profile in individuals without diabetes. Am J Clin Nutr. 2025 Feb;121(2):246-255. doi: 10.1016/j.ajcnut.2024.11.028. Epub 2024 Nov 28. PMID 39615596
- [Derived] Hjort A, Bergia RE, Vitale M, Costabile G, Giacco R, Riccardi G, Campbell WW, Landberg R. Low- versus High-Glycemic Index Mediterranean-Style Eating Patterns Improved Some Domains of Health-Related Quality of Life but Not Sleep in Adults at Risk for Type 2 Diabetes: The MEDGICarb Randomized Controlled Trial. J Nutr. 2024 Sep;154(9):2743-2751. doi: 10.1016/j.tjnut.2024.07.005. Epub 2024 Jul 14. PMID 39004223
- [Derived] Costabile G, Bergia RE, Vitale M, Hjorth T, Campbell W, Landberg R, Riccardi G, Giacco R. Effects on cardiovascular risk factors of a low- vs high-glycemic index Mediterranean diet in high cardiometabolic risk individuals: the MEDGI-Carb study. Eur J Clin Nutr. 2024 May;78(5):384-390. doi: 10.1038/s41430-024-01406-y. Epub 2024 Jan 24. PMID 38267533
- [Derived] Vitale M, Costabile G, Bergia RE, Hjorth T, Campbell WW, Landberg R, Riccardi G, Giacco R. The effects of Mediterranean diets with low or high glycemic index on plasma glucose and insulin profiles are different in adult men and women: Data from MEDGI-Carb randomized clinical trial. Clin Nutr. 2023 Oct;42(10):2022-2028. doi: 10.1016/j.clnu.2023.08.016. Epub 2023 Aug 25. PMID 37651979
- [Derived] Bergia RE 3rd, Biskup I, Giacco R, Costabile G, Gray S, Wright A, Vitale M, Campbell WW, Landberg R, Riccardi G. The MEDGICarb-Study: Design of a multi-center randomized controlled trial to determine the differential health-promoting effects of low- and high-glycemic index Mediterranean-style eating patterns. Contemp Clin Trials Commun. 2020 Aug 13;19:100640. doi: 10.1016/j.conctc.2020.100640. eCollection 2020 Sep. PMID 32885091